CLINICAL TRIAL: NCT07116265
Title: Long Term Clinical and Hemodynamic Follow-up of the Sutureless Perceval Bioprothesis
Brief Title: Perceval Aortic Bioprostheses : Durability Study.
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-MTP_2023_07_202301441
Record Dates: First submitted 2025-07-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Stenoses, Aortic Valve; Aortic Insufficiency; Aortic Diseases
Keywords: perceval; durability; degeneration; pacemaker
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency; Aortic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aortic valve replacement is one of the most commonly performed procedures in adult cardiac surgery in France.

Patients over the age of 65 most often receive a bioprosthetic aortic valve during an isolated aortic valve replacement or in combination with another cardiac surgery, which may extend the operative time.

The Perceval bioprosthesis has the advantage to reduce operative time due to its automatic deployment on a stent, which shortens the suturing time compared to other bioprostheses that require more sutures (sutureless valve).

In this retrospective, single-center, observational descriptive study, the investigators are conducting a follow-up of 193 patients operated on at the Montpellier University Hospital between January 2012 and January 2023, who received a Perceval aortic valve as part of routine annual follow-up, in order to assess the durability of this valve based on clinical and echocardiographic Valve Academic Research Consortium 3 (VARC-3) criteria.

DETAILED DESCRIPTION:
Exclusion Criteria :

Perceval bioprosthesis explanted during the same surgical procedure. History of aortic root surgery.

Primary Endpoint :

- Survival free from valve degeneration, according to VARC-3 criteria for structural or non-structural valve dysfunction.

Secondary endpoints :

* Freedom from aortic valve reintervention
* Freedom from SVD
* Freedom from permanent pacemaker implantation
* Freedom from stroke or transient ischemic attack
* Freedom from cardiac related rehospitalization
* Cardiac-specific mortality

Preoperative clinical data are collected via the DxCare electronic medical record system (including weight, height, medical history, and cardiovascular risk factors). Surgical data (type of procedure, operative time, outcomes at the end of surgery) are also extracted from the same software.

Follow-up Procedures :

Included patients are systematically scheduled for a cardiology follow-up consultation as part of routine annual postoperative care at the university hospital or in private practice. During this visit, they undergo a transthoracic echocardiography and a clinical assessment of their health status. These data are collected for analysis.

If patients are not followed up at the hospital and are considered lost to follow-up, their referring cardiologist will be contacted to obtain the most recent cardiological health data.

The annual follow-up echocardiography focuses on evaluating the hemodynamic parameters and durability of the bioprosthesis (presence or absence of pathological regurgitation, leaflet immobility, or thickening).

Clinical status is also assessed during the annual follow-up, including symptoms such as dyspnea, chest pain, and limitations in daily activities.

As part of standard follow-up, patients are contacted by phone and informed of the purpose of their scheduled visit to the Montpellier University Hospital.

For patients unable to attend an in-person consultation, a telephone interview is conducted to assess their clinical status, and their cardiologist is contacted to provide the most recent echocardiography report and clinical follow-up data. For patients who died before the beginning of the study, their trusted contact is approached to obtain clinical information regarding their medical history prior to death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe or non-severe aortic stenosis, symptomatic or asymptomatic, who received a rapidly deployed Perceval aortic bioprosthesis between January 1, 2012, and January 31, 2023, in the cardiac surgery department at Montpellier University Hospital.

Exclusion Criteria:

* Perceval bioprosthesis explanted during the same surgical procedure.
* History of aortic root surgery.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe or non-severe aortic disease, symptomatic or asymptomatic, who received a rapidly deployed Perceval aortic bioprosthesis between January 1, 2012, and January 31, 2023, in the cardiac surgery department at Montpellier University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
survival without Bioprosthetic Valve Failure | From enrollment to the last news (up to 130 months) or death

SECONDARY OUTCOMES:
Survival without reoperation | From enrollment to the last news (up to 130 months) or death
Survival without structural valve deterioration | From enrollment to the last news (up to 130 months) or death
survival without pacemaker implantation | From enrollment to the last news (up to 130 months) or death
survival without stroke | From enrollment to the last news (up to 130 months) or death
Survival without rehospitalization for cardiac origin | From enrollment to the last news (up to 130 months) or death
Survival without death for cardiac origin | From enrollment to the last news (up to 130 months) or death

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 31. Fischlein T, Meuris B, Hakim-Meibodi K, Misfeld M, Carrel T, Zembala M, et al. The sutureless aortic valve at 1 year: A large multicenter cohort study. JTCVS. (2016) ; 151(6):1617-1626.e4. 32. Fischlein T, Meuris B, Folliguet T, Hakim-Meibodi K, Misfeld M, Carrel T, et al. Midterm outcomes with a sutureless aortic bioprosthesis in a prospective multicenter cohort study. JTCVS. (2022) ; 164(6):1772-1780.e11. 35. Généreux P, Piazza N, Alu MC, Nazif T, Hahn RT, Pibarot P, et al. Valve Academic Research Consortium 3: Updated Endpoint Definitions for Aortic Valve Clinical Research. JACC. (2021) ; 77(21):2717-46.